CLINICAL TRIAL: NCT01813032
Title: Comparison of Vascular Function in Emergency Service Professionals
Acronym: FIRECOP
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: 11-SS-0085; PG/11/27/28842 (Other Grant/Funding Number: British Heart Foundation)
Record Dates: First submitted 2013-03-14; First posted 2013-03-18 (Estimated); Last update posted 2024-05-03 (Actual); Status verified 2013-03

CONDITIONS: Vascular Function; Atherothrombosis
Keywords: firefighters; police officers; emergency service professionals; myocardial infarction; endothelial function; thrombosis
MeSH Terms: conditions — Thrombosis; Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and urine.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Firefighters: 20 firefighters will attend for vascular assessments following a minimum of 48 hours off-duty.
  Interventions: Procedure: Forearm Vascular Study; Procedure: Badimon Chamber
- Police Officers: 20 police officers will attend for vascular assessments following a minimum of 48 hours off-duty.
  Interventions: Procedure: Forearm Vascular Study; Procedure: Badimon Chamber

INTERVENTIONS:
Procedure: Forearm Vascular Study — Forearm venous occlusion plethysmography to measure forearm blood flow during intra-arterial infusion of the vasodilators Verapamil (10-100 µg/min), bradykinin (100-1000 pmol/min), sodium nitroprusside (2-8 µg/min) and Acetylcholine (5-20 µg/min).
  Other Names: BK; SNP; ACh; VP
Procedure: Badimon Chamber — Ex-vivo assessment of thrombus formation using the Badimon Chamber

SUMMARY:
Emergency Service Professionals have an increased risk of death from heart attacks when compared to the general public. All the emergency professions share similar responsibilities such as emergency call-outs and shift work. Heart disease is the commonest cause of on-duty death amongst fire-fighters accounting for 45% and compared with 22% in police officers and 15% in the general population. The unique risk to fire-fighters is likely to reflect a combination of factors including extreme physical exertion, mental stress, heat and pollutant exposure.

In this study the investigators will assess healthy career fire-fighters and age-matched healthy police officer control subjects following a sedentary period. The investigators will take blood samples to measure platelet activity (platelets are the particles in blood that help blood clot) and will examine how blood clots outside of the body. The investigators will then perform studies placing small needles in the arm to assess how the blood vessels respond following these duties. The investigators hypothesise that fire-fighters do not have pre-existing impairment of heart, blood or blood vessel function as a cumulative effect of their occupation, but rather these are acute and transitory effects following distinct fire-fighter duties. We therefore expect similar results in both occupational groups.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking healthy firefighters

Exclusion Criteria:

* Current smoker
* History of lung or ischaemic heart disease
* Malignant arrhythmia
* Systolic blood pressure >190mmHg or <100mmHg
* Renal or hepatic dysfunction
* Previous history of blood dyscrasia
* Unable to tolerate the supine position
* Blood donation within the last 3 months
* Recent respiratory tract infection within the past 4 weeks
* Routine medication including aspirin and NSAIDs

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects will be healthy, non-smoking, whole-time firefighters working within Lothian and Borders Fire and Rescue Service and age- and sex-matched police officers who are also healthy and non-smokers working within Lothian and Borders Police Force.
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Forearm blood flow measured by venous occlusion plethysmography in response to infused vasodilators | following 48 hours off duty

SECONDARY OUTCOMES:
Ex-vivo thrombus formation using the Badimon chamber | following 48 hours off duty
Plasma t-PA and PAI concentrations following infusion of bradykinin | During forearm study, following 48 hours off duty

CONTACTS AND LOCATIONS:
Overall Officials: David E Newby, MD PhD, Study Chair — University of Edinburgh; Nicholas L Mills, MBChB PhD, Study Director — University of Edinburgh; Amanda L Hunter, MBChB, Principal Investigator — University of Edinburgh
Locations (1):
- Royal Infirmary of Edinburgh Clinical Research Facility, Edinburgh, United Kingdom